CLINICAL TRIAL: NCT01672086
Title: Active Surveillance Post-Approval Atudy of the Stelkast Surpass Acetabular System
Status: Terminated | Type: Observational
Why Stopped: Product is no longer being manufactured and marketed.
Sponsor: StelKast, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 344-01
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Survivorship and Long-term Safety and Effectiveness of the Stelkast Surpass Acetabular System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stelkast Surpass Patients
  Interventions: Device: Stelkast Surpass Acetabular System implant

INTERVENTIONS:
Device: Stelkast Surpass Acetabular System implant

SUMMARY:
The active surveillance post-approval study of the Stelkast Surpass Acetabular System is a retrospective, multi-center, single-arm study intended to collect data on the survivorship and long-term safety and effectiveness of the device.

DETAILED DESCRIPTION:
This active surveillance study is intended to evaluate the survivorship and long-term safety and effectiveness of the Stelkast Surpass Acetabular System. Neither the patient nor the surgeon are blinded to treatment. The study will compare the Surpass' survivorship to the survivorship observed in a historical control group established by a meta-analysis. The evaluation will be conducted for a period of ten years. These evaluations will be recorded through onsite visits and/or mailings sent to physicians requesting deidentified patient-level data for subjects implanted with the Surpass system.

ELIGIBILITY:
Inclusion Criteria:

* Primary hip arthroplasty
* Skeletal maturity
* Non-inflammatory degenerative joint disease such as osteoarthritis, avascular necrosis, congenital hip dysplasia, and traumatic arthritis

Exclusion Criteria:

* The Stelkast Surpass Acetabular System is contraindicated in patients with the following conditions: Overt or latent infection in or around the hip joint, insufficient bone stock to allow appropriate insertion and fixation of the prosthesis, insufficient soft tissue integrity to provide adequate stability, muscle laxity or inadequate soft tissue for proper function and healing, mental or neuromuscular disorders that do not allow control of the affected joint, revision hip arthroplasty, inflammatory hip joint disease, and neuropathic hip joint disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with the Stelkast Surpass Acetabular System at the participating siteswill be included in the evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2012-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Survivorship | 10 Years

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Allen, Study Director — MCRA
Locations (4):
- United States (4):
  - Gill Orthopedic Clinic, Charlotte, North Carolina
  - Mutschler Orthopedic Institute, Canonsburg, Pennsylvania
  - Premier Orthopedics and SPM Associates, Glen Mills, Pennsylvania
  - The Rothman Institute, Philadelphia, Pennsylvania